CLINICAL TRIAL: NCT02795533
Title: Changes in Physical, Cognitive and Emotional Function 5 and 10 Years After Aneurysmal Subarachnoid Hemorrhage (aSAH)
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tonje Haug Nordenmark, PhD, Oslo University Hospital
Other Study IDs: 2016/422
Record Dates: First submitted 2016-05-31; First posted 2016-06-10 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Cognitive function; Quality of Life
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical follow-up: As part of the regular follow-up of aSAH patients at Oslo University Hospital patients with as aSAH in 2011-2012 will be invited to a clinical interview, medical examination and neuropsychological test. Patients will also be asked to answer Quality of Life Questionnaires.
  Interventions: Behavioral: Clinical follow-up

INTERVENTIONS:
Behavioral: Clinical follow-up — All included patients will have a clinical follow-up consisting of:
  1. A medical examination
  2. Quality of life questionnaires
  3. Neuropsychological test
  All instruments have been translated into Norwegian and validated and tested in clinical practice.

SUMMARY:
The current study is a continuation of the study "Effect of early rehabilitation in patients with acute aSAH" which was approved by the Regional Committee for Medical Research Ethics, South-East Norway, archive number 2011/2189, Clinical Trials number 0925-0586 (Clinical Trials gov. identifier NCT01656317). The original study was a prospective, controlled, interventional study comprising patients managed at the neuro-intermediate ward following repair of a ruptured intracranial aneurysm in 2011-2012. 157 patients signed the informed consent form and were included in the study. Patients were assessed in the acute phase, as well as a 3 and 12 months post ictus. The main research goal of the present study will be to assess physical, cognitive and emotional function 5 and 10 years after aSAH in the 2011-2012 population. In addition we will also describe quality of life and work-status along with the time-course of recovery from the acute sage after aSAH to the chronic phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aSAH treated at Oslo University Hospital in 2011-2012
* Only patients with signed informed consent form and thereby included the project "Effect of early rehabilitation in patients with acute subarachnoid hemorrhage" (Regional Committee for Medical Research Ethics, South-East Norway, archive number 2011/2189, Clinical Trials number 0925-0586, Clinical Trials gov. identifier NCT01656317) will be asked to participate.

Exclusion criteria:

* Patients with aSAH treated at Oslo University Hospital in 2011-2012 who did not sign an informed consent form in the project "Effect of early rehabilitation in patients with acute subarachnoid hemorrhage" (Regional Committee for Medical Research Ethics, South-East Norway, archive number 2011/2189, Clinical Trials number 0925-0586, Clinical Trials gov. identifier NCT01656317)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for aSAH at Oslo University Hospital in 2011-2012
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
The Rivermead Post Concussion Symptom Questionnaire (RPQ) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Questionnaire

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Questionnaire
Fatigue Severity Scale (FSS) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Questionnaire
Mental Fatigue Scale (MFS) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Questionnaire
Behavioral Rating Inventory of Executive Function- Adult version (BRIEF-A) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Questionnaire
California Verbal Learning Test (CVLT) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test of verbal learning and memory
Color-Word interference test, Delis-Kaplan Test of Executive Function System | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test of executive functions
Digit span, Wechsler Adult Intelligence Scale-IV | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test of working memory
Mini Mental Status Examination (MMSE-NR3) | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test
Breif Visual Memory Test | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test of visual memory
Grooved Pegboard | Patients with an aSAH in 2011 will have their 5 years assessment in 2016 and 10 year assessment in 2021. Patients with an aSAH in 2012 will have their 5 year assessment in 2017 and 10 year assessment in 2022
  Test of motor skills

CONTACTS AND LOCATIONS:
Overall Officials: Tonje Haug Nordenmark, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Department of Physical medicine and rehabilitation, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No